CLINICAL TRIAL: NCT06001190
Title: The Influence of Oral Probiotic on the Vaginal Flora and Microenvironment Alteration in the Vaginosis Infection Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CORPG6M0171
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Probiotic, Human Papillomavirus Infection, Pap Smear, Microbiome
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotic intervention (Active Comparator): probiotic group with daily treatment
  Interventions: Dietary Supplement: probiotic:Lactobacillus crispatus
- placebo (Placebo Comparator): placebo-controlled with daily treatment
  Interventions: Dietary Supplement: probiotic:Lactobacillus crispatus

INTERVENTIONS:
Dietary Supplement: probiotic:Lactobacillus crispatus — We seek to observe that probiotic supplement(arm A) can improve vagina microbiome distribution by comapred to placebo group(arm B) in our study.

SUMMARY:
A single-blind, randomized, and probiotic-treatment including adult women with vaginitis and/or HPV positive. After oral probiotics, all participants will be followd-up cervical swabs and vaginal microbiome alteration till the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as vaginal viginitis
* willing to sign permit
* willing to regular follow up

Exclusion Criteria:

* Pregnant
* Virgin
* Severe cervix pathology CINII or CIN III
* Confirmed cervical cancer
* under long term antibiotics due to other physical condition

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
improvement alteration of vaginal microbiome | 3 months
  16s rRNA

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided